CLINICAL TRIAL: NCT02893540
Title: Capecitabine Metronomic Chemotherapy Versus Conventional Chemotherapy as Maintenance Treatment in Metastatic Colorectal Cancer
Brief Title: Metronomic Versus Conventional Chemotherapy in as Maintenance Treatment in mCRC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, MD, Ph.D, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH-Oncol-Metronomic
Record Dates: First submitted 2016-09-03; First posted 2016-09-08 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronomic (Experimental): accept capecitabine metronomic chemotherapy (500mg, twice per day, everyday)
  Interventions: Drug: Capecitabine
- Conventional (Active Comparator): accept capecitabine conventional chemotherapy (1000mg/m2, twice per day for 14 days, every 21 days)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — we are going to compare two maintenance treatment models with capecitabine in this study
  Other Names: Xeloda

SUMMARY:
The optimum regimen of maintenance treatment after first-line chemotherapy in patients with metastatic colorectal cancer (mCRC) is unknown. This study was designed to determine the efficacy and safety of maintenance treatment with capecitabine metronomic chemotherapy versus conventional chemotherapy.

DETAILED DESCRIPTION:
In this Prospective, open-label, randomised controlled trial, the investigators will recruit 250 mCRC patients who have finished 18 to 24 weeks first-line chemotherapy and disease evaluation is SD, PR or CR. Then, the patients will be randomised into two group. The experimental group, capecitabine metronomic chemotherapy versus capecitabine conventional chemotherapy as control group. These treatment regimens will be continued until progression, death, or an unacceptable adverse event.

The primary endpoint is progression-free survival (PFS). Secondary endpoints are overall survival (OS), quality of life (QOL) and toxic effects.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal cancer (in case of a single metastasis, histological or cytological proof of this lesion should be obtained);
* Distant metastases (patients with only local recurrence are not eligible);
* Unidimensionally measurable disease (> 1 cm on spiral CT scan or > 2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation;
* In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field.

Exclusion Criteria:

* Prior adjuvant treatment for stage II/III colorectal cancer ending within 6 months before the start of induction treatment;
* Any prior adjuvant treatment after resection of distant metastases;
* Previous systemic treatment for advanced disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
PFS1 | 4 months
  from randomizing to progression

SECONDARY OUTCOMES:
OS | 20 months
  from signing informed consent form to death
QOL | 20 months
  QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Wang, MD, Principal Investigator — Shanghai Rui Jin Hospital
Locations (1):
- Shanghai Rui Jin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simkens LH, van Tinteren H, May A, ten Tije AJ, Creemers GJ, Loosveld OJ, de Jongh FE, Erdkamp FL, Erjavec Z, van der Torren AM, Tol J, Braun HJ, Nieboer P, van der Hoeven JJ, Haasjes JG, Jansen RL, Wals J, Cats A, Derleyn VA, Honkoop AH, Mol L, Punt CJ, Koopman M. Maintenance treatment with capecitabine and bevacizumab in metastatic colorectal cancer (CAIRO3): a phase 3 randomised controlled trial of the Dutch Colorectal Cancer Group. Lancet. 2015 May 9;385(9980):1843-52. doi: 10.1016/S0140-6736(14)62004-3. Epub 2015 Apr 7. PMID 25862517
- [Background] Luo HY, Li YH, Wang W, Wang ZQ, Yuan X, Ma D, Wang FH, Zhang DS, Lin DR, Lin YC, Jia J, Hu XH, Peng JW, Xu RH. Single-agent capecitabine as maintenance therapy after induction of XELOX (or FOLFOX) in first-line treatment of metastatic colorectal cancer: randomized clinical trial of efficacy and safety. Ann Oncol. 2016 Jun;27(6):1074-1081. doi: 10.1093/annonc/mdw101. Epub 2016 Mar 2. PMID 26940686